CLINICAL TRIAL: NCT02681055
Title: An Open-Label Study To Evaluate The Efficacy, Safety, Tolerability and PK of MN-001 (Tipelukast) on HDL Function and Serum Triglyceride Levels in NASH and Non-Alcoholic Fatty Liver Disease (NAFLD) Subjects With Hypertriglyceridemia
Brief Title: Open-Label Study To Evaluate MN-001 on HDL & Triglyceride in NASH & NAFLD Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MN-001-NATG-201
Record Dates: First submitted 2016-02-05; First posted 2016-02-12 (Estimated); Results first posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Non-alcoholic Steatohepatitis; Hypertriglyceridemia; Non-alcoholic Fatty Liver Disease; Hypercholesterolemia
Keywords: NASH; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hypertriglyceridemia; Hypercholesterolemia | interventions — 4-(6-acetyl-3-(3-(4-acetyl-3-hydroxy-2-propylphenylthio)propoxy)-2-propylphenoxy)butyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label arm (Experimental): All 40 subjects will receive MN-001 for the first 4 weeks. At Week 4 subjects will increase their dosage frequency for remaining 8 weeks. Subjects will receive MN-001 for a total of 12 weeks.
  Interventions: Drug: MN-001

INTERVENTIONS:
Drug: MN-001 — MN-001 is a novel, orally bioavailable small molecule compound which demonstrates anti-inflammatory activity
  Other Names: tipelukast

SUMMARY:
This is a multi-center, proof-of-principle, open-label study designed to evaluate the efficacy, safety, and tolerability of MN-001 in non-alcoholic steatohepatitis (NASH) and Non-Alcoholic Fatty Liver Disease (NAFLD) subjects with hypertriglyceridemia.

DETAILED DESCRIPTION:
The study will consist a Screening Phase (up to 4 months) followed by a Treatment Phase (12 weeks), and a Follow-up visit (within 1 week after the last dose). A total of 40 male and female subjects ≥18 years of age are planned to be enrolled. During the Screening Phase, subjects will be assessed for study eligibility. After signing the informed consent form, the following assessments will be performed: medical history including review of prior and current medications, physical examination including height and body weight, waist circumference, vital signs and an electrocardiogram. Clinical labs, routine chemistries, hematology, coagulation profile, urinalysis and a serum pregnancy test will be collected as well as cytokeratin-18 (CK-18), a biomarker for NASH diagnosis. An alcohol consumption questionnaire will be administered and a MRI scan of the liver will be performed. Serum fibrosis markers, the Fib-4 index (age, AST, ALT, PLT) and NAFLD fibrosis score (age, BMI, AST/ALT ratio, IFG/DM, PLT, Albumin) will be calculated.

ELIGIBILITY:
INCLUSION CRITERIA:

* Written informed consent is obtained and willing and able to comply with the protocol in the opinion of the Investigator.
* Male or female subjects ≥ 18 years of age
* Histologically proven NASH (NAFLD activity score of 3 or greater with at least 1 point being ballooning) based on liver biopsy performed within the last 36 months or abdominal ultrasound confirmation of non-alcoholic fatty liver disease (NAFLD)
* Fasting serum triglyceride level > 150 mg/dL (confirmed at screening)
* Serum ALT, AST, ALP and total bilirubin levels at Screening (- 120 days to -30 days) and Lab Visit values (- 1 week ± 5 days) are stable or changes at the Lab visit are < 20% of the values from Screening.
* BMI ≤ 45 kg/m2
* Subjects on the following medications can be enrolled if these medications are necessary, cannot be stopped, and the dose has been stable for 4 months or more prior to baseline:

  * Stable doses of anti-diabetic medications
  * Stable doses of fibrates, statins, niacin, ezetimibe.
  * Stable doses of Vitamin E for at least 8 weeks
* Less than 21 units of alcohol/week for men and 14 units of alcohol/week for women over a 2-year time frame
* Females of child-bearing potential must have a negative serum ß-hCG at screening and must be willing to use appropriate contraception (as defined by the investigator) for the duration of study treatment and 30 days after the last dose of study treatment.
* Males should practice contraception as follows: condom use and contraception by female partner.
* Subject is in good physical health on the basis of medical history, physical examination, and laboratory screening, as defined by the investigator.
* Subject is willing and able to comply with the protocol assessments and visits, in the opinion of the study nurse/coordinator and the Investigator.

EXCLUSION CRITERIA:

* Diagnosis of other known cause of liver disease (autoimmune, viral, genetic, drug- or alcohol-induced, or storage disease)
* Decompensated or severe liver disease defined by one or more of the following:
* biopsy-proven cirrhosis
* INR >1.5
* Total bilirubin (TBL) > 1.5 x ULN, or > 2 x ULN for unconjugated bilirubin
* serum albumin <2.8 g/dL
* ALT or AST > 10 x ULN
* evidence of portal hypertension including splenomegaly, ascites, encephalopathy and/or esophageal varices
* Current diagnosis of hepatocellular carcinoma (HCC) or suspicion of HCC clinically or on ultrasound
* Uncontrolled diabetes mellitus Type 2
* History of bariatric surgery
* Greater than 10-pound weight gain or loss in the last 6 months
* Clinically significant cardiovascular/cerebrovascular disease, including myocardial infarct within last 6 months, coronary artery intervention, coronary artery bypass, unstable ischemic heart disease, heart failure class III or IV, angina or cerebral vascular accident.
* Resting pulse < 50 bpm, SA or AV block, uncontrolled hypertension, or QTcF > 450 ms
* History of stomach or intestinal surgery or any other condition that could interfere with or is judged by the Investigator to interfere with absorption, distribution, metabolism, or excretion of study drug.
* Any significant laboratory abnormality which, in the opinion of the Investigator, may put the subject at risk
* History of malignancy < 5 years prior to signing the informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* History of HIV (human immunodeficiency virus), HBV, HCV (cured HCV is not excluded), EBV CMV or other active infection.
* Currently has a clinically significant medical condition including the following: neurological, psychiatric, metabolic, immunologic, hematological, pulmonary, cardiovascular (including uncontrolled hypertension), gastrointestinal, urological disorder, or central nervous system (CNS) infection that would pose a risk to the subject if they were to participate in the study or that might confound the results of the study. Note: Active medical conditions that are minor or well-controlled are not exclusionary if, in the judgment of the Investigator, they do not affect risk to the subject or the study results. In cases in which the impact of the condition upon risk to the subject or study results is unclear, the Medical Safety Monitor should be consulted.
* CYP2C8 substrates with a narrow therapeutic index (e.g., paclitaxel) within 15 days prior to study and throughout the study are prohibited.
* CYP2C9 substrate with narrow therapeutic index (e.g., phenytoin, S-warfarin, tolbutamide) within 15 days prior to study and throughout the study are prohibited.
* Macrolide or quinolone class antibiotics within 15 days of Screening Visit and throughout the study are prohibited.
* Steroids within 30 days prior to study drug dosing and throughout the study unless administered for a short term treatment course during the study are prohibited.
* History of alcohol or substance abuse (DSM-IV-TR criteria) within 3 months prior to screening or alcohol or substance dependence (DSM-IV-TR criteria) within 12 months prior to screening. The only exceptions include caffeine or nicotine abuse/dependence.
* Poor peripheral venous access that will limit the ability to draw blood as judged by the Investigator.
* Currently participating, or has participated in, a study with an investigational or marketed compound or device within 3 months prior to signing the informed consent.
* Unable to cooperate with any study procedures, unlikely to adhere to the study procedures and keep appointments, in the opinion of the Investigator, or was planning to relocate during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuko Matsuda, MD PhD MPH, Study Chair — MediciNova
Locations (3):
- United States (3):
  - Southern California Research Center, Coronado, California
  - Scripps Research, La Jolla, California
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Arm: All subjects will take MN-001 250 mg once a day for the first 4 weeks. After 4 weeks of MN-001 250 mg once a day, all subjects will take MN-001 250 mg twice a day for the remaining 8 weeks of the treatment phase. Subjects will receive MN-001 for a total of 12 weeks.
Period: Weeks 1-4
Arm/Group | Open Label Arm
Started | 19
Completed | 19
Not Completed | 0
Period: Weeks 5-12
Arm/Group | Open Label Arm
Started | 19
Completed | 18
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Open Label Arm: All 19 subjects will receive MN-001 for the first 4 weeks. At Week 4 subjects will increase their dosage frequency for remaining 8 weeks. Subjects will receive MN-001 for a total of 12 weeks.
  MN-001: MN-001 is a novel, orally bioavailable small molecule compound which demonstrates anti-inflammatory activity
Arm/Group | Open Label Arm
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 54.6 [27 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline at 12 Weeks of MN-001 Treatment on Cholesterol Efflux Capacity
Description: Change from baseline to 12 weeks of MN-001 on Cholesterol Efflux Capacity (CEC) in NAFLD subjects with hypertriglyceridemia. CEC, a key step in reverse cholesterol transport, was inversely associated with the incidence of cardiovascular events and is considered to be a new biomarker to assess cardiovascular risk. Cholesterol efflux was calculated as the percent of cholesterol removed from the cells and appearing in the culture medium normalized to a reference serum pool. The ability of serum HDL to remove cholesterol from cultured cells was assessed as an in vitro method to evaluate functional changes in HDL mediated by changes due to MN-001 treatment.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of cholesterol
Arm/Group | Open Label Arm
Number analyzed (Participants) | 19
percentage of cholesterol | -0.013 (0.1022)

2. Primary Outcome: Mean Change From Baseline to Week 8 on Triglyceride Levels After 8 Weeks MN-001 Treatment
Description: Change from baseline to 8 weeks of MN-001 on serum triglyceride levels in NASH subjects with hypertriglyceridemia
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open Label Arm
Number analyzed (Participants) | 19
mg/dL | -21.67 (27.89)

3. Secondary Outcome: Number of Treatment-emergent Adverse Events
Description: Safety and tolerability of MN-001 by assessing the number of subjects who experienced treatment-emergent adverse events. A treatment-emergent adverse event is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with the trial intervention.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 13
Population: Safety population
Measure: Number; unit: number of adverse events
Groups:
- Open Label Arm: All 19 subjects will receive MN-001 for the first 4 weeks. At Week 5, subjects will increase their dosage frequency for remaining 8 weeks. Subjects will receive MN-001 for a total of 12 weeks.
  MN-001: MN-001 is a novel, orally bioavailable small molecule compound which demonstrates anti-inflammatory activity
Arm/Group | Open Label Arm
Number analyzed (Participants) | 19
number of adverse events
  All-cause mortality | 0
  serious adverse events | 0
  adverse events | 18

4. Secondary Outcome: Mean Plasma Concentration of MN-001 and MN-002 (Metabolite) After a Single Dose of MN-001 in Six Subjects
Description: Mean plasma concentration of of MN-001 and its metabolite, MN-002, after a single 250 mg oral dose of MN-001 in nonalcoholic steatohepatitis and nonalcoholic fatty liver disease patients.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Open Label Arm
Number analyzed (Participants) | 6
mcg/mL
  Mean plasma concentration of MN-001 after a single dose of MN-001 250 mg | 0.434 (0.205)
  Mean plasma concentration of MN-002 after a single dose of MN-001 250 mg | 3.44 (2.40)

5. Secondary Outcome: Mean Serum Lipids From Baseline to Week 8
Description: Mean change from baseline to week 8 on total cholesterol, high-density lipoproteins, low-density lipoproteins
Time Frame: Baseline, Week 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open Label Arm
Number analyzed (Participants) | 19
mg/dL
  Total cholesterol | -15.2 (41.34)
  high-density lipoproteins | 3.2 (7.61)
  low-density lipoproteins | -13.7 (55.31)

6. Secondary Outcome: Mean Change in Liver Enzymes From Baseline to Week 8
Description: Measure the effect of MN-001/002 on alanine aminotransferase (ALT) and aspartate aminotransferase (AST) mean change from Baseline to Week 8
Time Frame: Baseline, Week 8
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Open Label Arm
Number analyzed (Participants) | 19
U/L
  alanine aminotransferase | -5.7 (22.79)
  aspartate aminotransferase | 1.2 (22.7)

7. Secondary Outcome: Measure the Effect of MN-001/002 on Percentage of Fat in the Liver
Description: To measure the effect of MN-001/002 on percentage of fat in the liver by MRI mean change from baseline to Week 12
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: percentage of fat in liver
Arm/Group | Open Label Arm
Number analyzed (Participants) | 19
percentage of fat in liver | 0.64 (5.54)

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | Open Label Arm
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 10/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Arm (N=19)
diarrhea (Gastrointestinal disorders) | 2 (2)
constipation (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
ear infection (Infections and infestations) | 1 (1)
nasopharyngitis (Infections and infestations) | 1 (1)
alanine aminotransferase increased (Investigations) | 1 (1)
aspartate aminotransferase increased (Investigations) | 1 (1)
heart rate increased (Investigations) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
hypoaesthesia (Nervous system disorders) | 1 (1)
paraesthesia (Nervous system disorders) | 1 (1)
bundle branch block left (Cardiac disorders) | 1 (1)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1)
phlebitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT02681055/Prot_SAP_ICF_001.pdf